CLINICAL TRIAL: NCT01984476
Title: Impact of Age on Cardiovascular, Cerebrovascular and Cognitive Health in Spinal Cord Injury
Status: Completed | Type: Observational
Sponsor: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Jill M. Wecht, Ed.D., Research Health Scientist, James J. Peters Veterans Affairs Medical Center
Other Study IDs: WEC-13-042
Record Dates: First submitted 2013-11-08; First posted 2013-11-14 (Estimated); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: Spinal Cord Injury
Keywords: spinal cord injury; autonomic dysreflexia; baroreceptor integrity; sympathetic integrity; vagal integrity; autonomic integrity; arterial stiffness; cognitive function; traumatic brain injury; cerebral blood flow; white matter hyperintensities; cerebral vascular resistance index
MeSH Terms: conditions — Spinal Cord Injuries; Autonomic Dysreflexia; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Older Able-Bodied Controls: Subjects must be between the age of 55 and 65 years old, be English-literate and able to provide informed consent. They must score at least 20/60 minimum acuity in their worst eye on the Snell Eye Exam, and score at least 24 on the Montreal Cognitive Assessment. Subjects MUST NOT HAVE: an acute illness or infection, history of stroke, recent illicit drug abuse (<6 months), controlled or uncontrolled hypertension or diabetes mellitus, history of epilepsy or other seizure disorder, history of Traumatic Brain Injury (as determined by TBI screening tool), any significant history of neurological disease/disorder, and diagnosis of a psychiatric disorder such as post-traumatic stress disorder, schizophrenia or bipolar disorder.
- Spinal Cord Injured: Subjects must be between the age of 25 and 49 years old, be English-literate and able to provide informed consent. They must be injured between 5 to 10 years, level of injury between C1-T12, non-ambulatory (wheelchair dependent), and AIS grade of A or B. They must score at least 20/60 minimum acuity in their worst eye on the Snell Eye Exam, and score at least 24 on the Montreal Cognitive Assessment. Subjects MUST NOT HAVE: an acute illness or infection, history of stroke, recent illicit drug abuse (<6 months), controlled or uncontrolled hypertension or diabetes mellitus, history of epilepsy or other seizure disorder, history of Traumatic Brain Injury (as determined by TBI screening tool), any significant history of neurological disease/disorder, and diagnosis of a psychiatric disorder such as post-traumatic stress disorder, schizophrenia or bipolar disorder.
- Age-Matched Able-Bodied Controls: Subjects must be between the age of 25 and 49 years old, be English-literate and able to provide informed consent. They must score at least 20/60 minimum acuity in their worst eye on the Snell Eye Exam, and score at least 24 on the Montreal Cognitive Assessment. Subjects MUST NOT HAVE: an acute illness or infection, history of stroke, recent illicit drug abuse (<6 months), controlled or uncontrolled hypertension or diabetes mellitus, history of epilepsy or other seizure disorder, history of Traumatic Brain Injury (as determined by TBI screening tool), any significant history of neurological disease/disorder, and diagnosis of a psychiatric disorder such as post-traumatic stress disorder, schizophrenia or bipolar disorder.

SUMMARY:
As the spinal cord injured population ages, these individuals are being exposed to an increased prevalence of age-associated diseases, which coupled with the secondary complications of the injury may contribute to the reduced life expectancies. Decentralized autonomic regulation in persons with SCI results in a multitude of cardiovascular changes, which may contribute to accelerated aging. Adverse cardiovascular changes may have deleterious effects on cerebral blood flow dynamics and an increase in cerebral vascular resistance index in individuals with SCI during cognitive testing. Deficits in memory and processing speed in individuals with SCI may relate to cardiovascular and cerebrovascular dysfunction. Identifying the associations between healthy aging versus premature or accelerated aging in organ system function in the SCI population is an important first step towards prevention and amelioration of these changes. Therefore the study objectives are to compare, among individuals with SCI, age-matched non-SCI and older non-SCI individuals arterial stiffness and cerebral vascular resistance index; memory, processing speed, and executive function; and volume of white matter hyperintensities. 60 individuals with SCI, 30 age-matched non-SCI controls, and 20 older non-SCI controls will be recruited for this study. All potential subjects will undergo a two-part screening process which consists of an initial screening via telephone and a detailed, in-person screening. Eligible subjects will be invited to participate in a 4 hour laboratory visit during which their arterial stiffness, blood pressure, heart rate, respiration rate and, blood flow to the brain will be monitored at rest and during a comprehensive series of cognitive tests. A subset of the participants will be asked to take part in an MRI brain imaging session: 40 persons with SCI, 10 age-matched non-SCI and 10 older non-SCI. Eligible subjects will be asked to participate in a 1 hour MRI/functional magnetic resonance imaging(fMRI) session.

We hypothesize that arterial stiffness and cerebral vascular resistance index will be increased in the SCI group compared to the age-matched non-SCI but will be comparable to the older non-SCI groups. In addition, we hypothesize that the prevalence of mild to moderate cognitive impairments in memory, processing speed, and executive function will be increased in the SCI individuals compared to the age-matched non-SCI but will be comparable to the older non-SCI individuals.

DETAILED DESCRIPTION:
The cognitive test battery will consists of the tests listed below, administered in the order given.

1. Digit Span
2. California Verbal Learning Test
3. Symbol Digit Modalities Test
4. Letter Number Sequencing
5. California Verbal Learning Test Delay
6. Paced Auditory Serial Addition Test
7. D-KEFS Verbal Fluency
8. D-KEFS Color-Word
9. WASI Vocabulary
10. WASI Matrix Reasoning

ELIGIBILITY:
Inclusion Criteria:

SCI

* Between the ages of 25 and 49 years old
* Duration of injury must be between 5 and 10 years
* AIS grade of A or B
* Non-ambulatory (wheelchair dependent)
* At least 20/60 minimum acuity in worst eye on the Snell Eye Exam
* A score ≥24 on the Montreal Cognitive Assessment
* English literate
* Able to provide informed consent

Age-matched non-SCI

* Between the ages of 25 and 49 years old
* At least 20/60 minimum acuity in worst eye on the Snell Eye Exam
* A score ≥24 on the Montreal Cognitive Assessment
* English literate
* Able to provide informed consent

Older non-SCI

* Between the ages of 55 and 65 years old
* At least 20/60 minimum acuity in worst eye on the Snell Eye Exam
* A score ≥24 on the Montreal Cognitive Assessment
* English literate
* Able to provide informed consent

Exclusion Criteria:

* Acute illness or infection
* Documented history of:
* Controlled or uncontrolled hypertension or Diabetes mellitus
* Recent illicit drug abuse (from medical chart, within the past 6-months)
* Epilepsy or seizures
* Neurodegenerative disease including Alzheimer's disease, Parkinson's disease, Dementia, Stroke, Multiple sclerosis
* Severe TBI (identified by TBI screening tool)
* Any significant history of psychiatric disease/disorders:
* Post-traumatic stress disorder
* schizophrenia
* Bipolar disease
* Substance abuse or dependence within the past 6 months

MRI has additional exclusion:

* Subject has been informed that it is medically unsafe to receive a regular MRI as part of my medical care
* Pregnant
* Right handed
* Prone to claustrophobia
* Metal in body including:
* metal fragments or pieces in subject's eye or any other part of body
* brain stimulators
* pacemakers, or other implanted electrical devices or pumps
* aneurysm clips
* metallic prostheses (including metal pins and rods, heart valves)
* internal hearing aids
* permanent eyeliner
* shrapnel fragments
* piercing that cannot be taken out

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 60 subjects with SCI, 30 age-matched non-SCI controls and 20 older non-SCI controls will be recruited from out-patient clinics at Kessler Institute for Rehabilitation. This includes subjects who have completed various protocols in the Cardiovascular autonomic testing laboratory or patients referred by their physicians following routine physical examinations. Physicians will be informed of the inclusion and exclusion criteria for this study and will be able to provide us with the assurance that the patient is an appropriate candidate for the study and that he/she was willing to speak with the study coordinators.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2013-07; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Arterial Stiffness | Up to 2 years
  To determine the difference in arterial stiffness among individuals with SCI to age-matched non-SCI and older non-SCI.
Cerebral Vascular Resistance Index | Up to 2 years
  To determine the difference in cerebral vascular resistance index among individuals with SCI to age-matched non-SCI and older non-SCI.

SECONDARY OUTCOMES:
Performance on Cognition Battery Tests | Up to 2 years
  To compare memory, processing speed, and executive function among individuals with SCI to age-matched non-SCI and older non-SCI.

OTHER OUTCOMES:
Volume of White Matter Hyperintensities | Up to 2 years
  To determine the difference in volume of white matter hyperintensities among individuals with SCI to age-matched non-SCI and older non-SCI.

CONTACTS AND LOCATIONS:
Overall Officials: Jill M Wecht, EdD, Principal Investigator — JJPVAMC
Locations (1):
- Kessler Foundation Research Center, West Orange, New Jersey, United States